CLINICAL TRIAL: NCT00544674
Title: A Phase II, Multi-Center, Open-Label, Trial of PR104 in Treatment Naive and Sensitive-relapse Small Cell Lung Cancer
Brief Title: PR104 in Treating Patients With Previously Untreated or Relapsed Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to discovery of new mechanism of activation.
Sponsor: Proacta, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR104-2001; PROACTA-PR-104-2001
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — PR-104; fluoromisonidazole

ARMS (1):
- PR104 (Experimental): PR104 will be administered once every 21 days by IV
  Interventions: Drug: PR104; Other: F-18-fluoromisonidazole

INTERVENTIONS:
Drug: PR104 — administered at a dose of 1100 mg/m^2 by intravenous infusion over 1 hour and repeated every three weeks
  Other Names: PR-104
Other: F-18-fluoromisonidazole — administered intravenously prior to PET scan
  Other Names: FMISO

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as PR-104, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well PR-104 works in treating patients with previously untreated or relapsed small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the response rate of PR-104 in patients with treatment-naive or sensitive-relapse small cell lung cancer.
* Evaluate safety of this drug in these patients. Secondary
* Evaluate survival of these patients.
* Evaluate progression-free survival of these patients.
* Evaluate time to progression in these patients.
* Assess the pharmacokinetics (PK) of PR-104 and its alcohol metabolite.
* Estimate the rate of hypoxia using 18F-fluoromisonidazole (FMISO) positron emission topography (PET) imaging.
* Collect plasma samples for assessment of potential biomarkers of tumor hypoxia.

OUTLINE: This is a multicenter study. Patients are stratified according to disease type (treatment-naive vs sensitive-relapse).

Patients receive PR-104 intravenously (IV) over 1 hour on day 1. Treatment repeats every 21 days for up to 4 courses (for treatment-naive patients) or in the absence of disease progression or unacceptable toxicity (for sensitive-relapse patients).

PK studies are performed during course 1 and after course 3. Blood is collected at baseline, during course 1, and at study completion for biomarker studies of tumor hypoxia (plasma proteins). Patients also undergo FMISO PET and fludeoxyglucose F18 (FDG) PET scans at baseline and after the second course of study therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically or cytologically confirmed small cell lung cancer (SCLC)
* If patient is treatment-naive, then they must have extensive disease
* If patients are not treatment-naive, then they must be classified as sensitive-relapse with either extensive disease or limited disease

  * Sensitive-relapse defined as disease that responded to first-line chemotherapy and relapsed more than 90 days following the last dose of first-line chemotherapy
  * Limited disease SCLC defined as disease confined to the hemithorax of origin, mediastinum, and/or ipsilateral supraclavicular lymph nodes, which could be encompassed within a tolerable radiotherapy port
  * Extensive disease defined as disease that does not fit the definition of limited disease as defined above
* Measurable or evaluable disease

Exclusion criteria:

* Active central nervous system (CNS) metastases, defined as metastases to the CNS (symptomatic or non-symptomatic) that requires immediate treatment or that are likely to require treatment in the following 6 weeks
* Medical conditions requiring urgent intervention, including any of the following:

  * Superior vena cava syndrome
  * Lobar obstruction
  * Spinal cord compression
  * Liver metastases involving greater than one-third of the liver

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (no red blood cell transfusions allowed)
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN (if liver metastases are present) or ≤ 2 x ULN (if liver metastases are absent)
* Serum creatinine ≤ 1.5 x ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 30 days after completion of study treatment

Exclusion criteria:

* Prior or concurrent malignancies, except for adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or localized low-grade prostate cancer
* Hyponatremia (< 130 mmol/L)
* Evidence of a significant medical disorder or laboratory finding that, in the opinion of the investigator, compromises the patient's safety during study participation, including any of the following:

  * Uncontrolled infection or infection requiring a concurrent parenteral antibiotic
  * Uncontrolled diabetes
  * Congestive heart failure
  * Myocardial infarction within the past 6 months
  * Chronic renal disease
  * Coagulopathy (excluding prophylactic anticoagulation)
* Known human immunodeficiency virus (HIV) positivity, hepatitis B surface antigen-positivity, or hepatitis C positivity with abnormal liver function tests

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* See Disease Characteristics
* No concurrent prophylactic growth factors (filgrastim [G-CSF] or sargramostim [GM-CSF]) during course 1 of study treatment

Exclusion criteria:

* More than one prior chemotherapy regimen for SCLC
* Less than 24 hours from any prior radiotherapy or the likelihood of toxicity from prior radiotherapy
* Radiotherapy to > 25% of the bone marrow within the past 4 weeks
* Less than four weeks since major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Arizona Clinical Research Center, Incorporated, Tucson, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Pacific Shores Medical Group - Long Beach, Long Beach, California
  - Stanford Cancer Center, Stanford, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Welborn Clinic, Evansville, Indiana
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Kentuckiana Cancer Institute, PLLC, Louisville, Kentucky
  - Purchase Cancer Group - Paducah, Paducah, Kentucky
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Cancer and Blood Specialists of Nevada - Henderson, Henderson, Nevada
  - Gabrail Cancer Center - Canton Office, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital Cancer Treatment Center, Cincinnati, Ohio
  - Peninsula Cancer Institute - Newport News Office, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- PR104: Subjects will receive 1100 mg/m^2 PR-104 intravenously once every 21 days (one cycle). In addition, subjects will undergo positron emission topography (PET) imaging with F-18-Fluoro Misonidazole (FMISO) for the assessment of hypoxia and with F-18-Fluorodeoxyglucose (FDG) for the assessment of glucose metabolism.
Period: Overall Study
Arm/Group | PR104
Started | 5 (1 subject registered and expired prior to dosing)
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- PR104: 1100 mg/m^2 PR104 by IV over one hour every three weeks
Arm/Group | PR104
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete or Partial)
Time Frame: From registration until disease progression/recurrence
Reporting Status: Not Posted
Measure: Number; unit: participants

2. Secondary Outcome: Survival
Time Frame: Every 3 months for 2 years after discontinuation
Reporting Status: Not Posted

3. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is the time (days) from date of registration to date of first observed disease progression (radiological or clinical, whichever was earlier) or death due to any cause, if death occurred before progression was documented.
Time Frame: Tumor measurements and assessments based on Response Evaluation Criteria In Solid Tumors (RECIST) criteria were performed 6 weeks after first dose and as dictated by subject's malignancy
Reporting Status: Not Posted

4. Secondary Outcome: Time to Progression
Description: Time to progression (TTP) was defined as the time from date of registration to radiological progression / recurrence. Subjects without progression at the time of analysis were censored at their last date of tumor evaluation.
Time Frame: From registration of the first subject until radiological progression or recurrence whichever came first
Reporting Status: Not Posted

5. Primary Outcome: Safety and Tolerability: the Number of Subjects Experiencing a Serious Adverse Events
Description: The number of participants with at least one Serious Adverse Event was measured.
Time Frame: 30 days following the last administration of study treatment
Measure: Number; unit: participants
Arm/Group | PR104
Number analyzed (Participants) | 4
participants | 2

6. Secondary Outcome: Pharmacokinetics
Time Frame: Days 1 and 2 of Cycles 1 and 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | PR104
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PR104 (N=4)
Vomiting (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PR104 (N=4)
Fatigue (General disorders) | 2
Chest pain (General disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Weight decreased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
Decision to close study early based on new data showing that PR104A could also be activated under oxic conditions in tumors that express high levels of AKR1C3. SCLC does not express meaningful levels of the enzyme aldo keto reductase 1C3 (AKR1C3).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Single site data may be published/presented prior to the publication of multi-center data from overall study if agreed to by the sponsor in writing, or 12 months have elapsed following termination or completion of the study, whichever comes first.